CLINICAL TRIAL: NCT05893017
Title: Comparison of the Effects of Different Treatment Modalities on Pain, Quality of Life, and Musculoskeletal System in Individuals with Knee Osteoarthritis
Brief Title: Comparison of the Effects of Different Treatment Modalities in Individuals with Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fatih Erbahceci, Prof. Dr. / Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E-68869993-511.06-765176
Record Dates: First submitted 2023-05-30; First posted 2023-06-07 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-02

CONDITIONS: Gonarthrosis; Primary
Keywords: Gonarthrosis; Virtual Reality Exercises; Valgus Orthosis; Kinesiotaping
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Virtual Reality Exercises (Experimental): Virtual Reality Exercises will be applied
  Interventions: Other: Virtual Reality Exercises
- Virtual Reality Exercises and Kinesiotaping (Experimental): Virtual Reality Exercises and Kinesio taping for quadriceps and hamstring muscles will be applied
  Interventions: Other: Virtual Reality Exercises and Kinesiotaping
- Virtual Reality Exercises and Valgus Orthoses (Experimental): Virtual Reality Exercises and Valgus Orthoses will be applied.
  Interventions: Other: Virtual Reality Exercises and Valgus Orthoses

INTERVENTIONS:
Other: Virtual Reality Exercises — Virtual Reality Exercises will be apply for muscle strengthening
  Arms: Virtual Reality Exercises
Other: Virtual Reality Exercises and Kinesiotaping — Virtual Reality Exercises will be apply for muscle strengthening, Kinesiotaping will be applied at Quadriceps muscle and Hamstring muscle
  Arms: Virtual Reality Exercises and Kinesiotaping
Other: Virtual Reality Exercises and Valgus Orthoses — Virtual Reality Exercises will be apply for muscle strengthening, Orthoses is for correction at knee alignment
  Arms: Virtual Reality Exercises and Valgus Orthoses

SUMMARY:
Knee osteoarthritis (gonarthrosis) is one of the most common types of osteoarthritis. It is a degenerative joint disorder characterized by pain, muscle weakness, and functional loss. There have been no studies comparing the effects of conservative treatment approaches such as virtual reality exercises, orthoses, and kinesio taping. Therefore, the aim of this current study is to compare the effectiveness of virtual reality exercises alone and in combination with orthotic approach and kinesio taping in individuals with knee osteoarthritis. The participants included in the study will be randomly divided into three groups. The first group will receive virtual reality exercises, the second group will receive virtual reality exercises along with valgus orthosis, and the third group will receive virtual reality exercises combined with kinesio taping treatment. The interventions will be applied three times a week for eight weeks. Evaluations will be repeated before and after the exercise therapy. The evaluations will include pain assessment using the Visual Analog Scale (VAS), muscle strength measured by hand dynamometer, balance assessed by the Berg Balance Scale, proprioception measured by stabilizer and inclinometer, joint range of motion measured by goniometer, functional status evaluated by the WOMAC scale, lower extremity length measured by tape measure, walking speed assessed by the 10-Meter Walk Test (10 MWT), quality of life measured by the SF-36 questionnaire, kinesiophobia evaluated by the Tampa Scale for Kinesiophobia, architectural features of the quadriceps femoris muscle assessed by ultrasound imaging, knee OA score measured by the Knee Injury and Osteoarthritis Outcome Score (KOOS), and medial compartment distance of the knee calculated and recorded using computer-aided analysis on anteroposterior radiographs.

DETAILED DESCRIPTION:
The patients to be evaluated in this study are those who were diagnosed with gonarthrosis and met the inclusion criteria. The study will be conducted with volunteer patients who accepted the voluntary consent form.

After the power analysis made in our research, at least 20 individuals in each group with 80% power and 0.05 margin of error.

It was found that a total of 60 individuals were required to participate. Demographic and clinical data of the patients to be included in the study will be obtained.

The patients will be randomized with the help of a computer program (www.randomizer.org) and divided into 3 groups. It will be formed by the patient group who received the Group-I Virtual Reality Exercises training. In addition to Group-II Virtual Reality Exercises training, it will be created by patients using valgus orthosis. Group-III will be formed by patients who receive kinesio taping treatments in addition to virtual reality exercises training. Virtual reality exercises will be applied with the help of Wii-Fit Balance Board (Nintendo of America Inc, Redmond, WA).

Virtual reality exercises are planned 3 times a week for 8 weeks, each session approximately 20-30 minutes and each game 3 repetitions. Balance games and yoga postures within the equipment will be used. "Ski Slalom and Table Tilt" are balance games, "Tree" and "Chair" are yoga posture poses.

Ski Slalom: Includes lateral weight transfer. The game can be played with squat position and weight transfer to the left and right.

Table Tilt: It aims to improve balance in many ways. The game can be played by transferring weight back and forth on the platform.

Tree pose: It is used to improve postural control. Chair pose: It is used to improve postural control. Tree stance pose and Chair stance pose create abduction moment in the hip and abduction moment in the knee. Low to moderate gonarthrosis of the hip abduction moment It has been reported that it will reduce the load on the medial compartment in patients.

Valgus orthosis; reducing the overload in the medial compartment of the knee showing varum alignment and it aims to increase the function. Increased activity and decreased pain may delay the need for surgery.

Kinesio taping; It will be applied to the quadriceps femoris and hamstring muscles of the patients as recommended by Kenzo Kase. For the quadriceps femoris muscle, the patient should be in the supine position with the knees straight. Y shaped tape will be used. The tape will be applied 5 cm below the SIAS with 25% tension, when it comes to the patella, it will be Y-shaped, starting from the proximal of the patella without tension by flexing the knee a little, and turning around it, and the taping will be finished in the inferior of the patella. Y-shaped tape will be used for hamsting muscle application. For taping, the patient should be standing and leaning forward from the trunk. The band will start from the ischial tuberosity and come to the back of the knee and will end medial and lateral to the knee.

Kinesio tape application will be applied immediately after the end of the virtual reality exercises session. Taping will be done 3 times a week for 8 weeks.

VAS: One of the most common problems in gonarthrosis is pain. Pain assessment will be done with Visual Analogue Scale (VAS). VAS; It is used to digitize the severity of pain that cannot be measured numerically. The two end definitions (0: No pain, 10: Unbearable pain) are written on the two ends of the 10-centimeter scale and the patient is asked to mark where his or her pain is in the scale.

Measurement of Knee Extension Muscle Strength: In order to measure muscle strength, methods such as manual muscle testing, isokinetic and isometric dynamometer or hand-held dynamometer (HHD) are used in the clinic.

Proprioceptive Force Sense Evaluation: It will be evaluated with a pressurized biofeedback device. They are asked to contract and hold for 5 seconds. The highest value read from the device during contractions of the patients is recorded in mmHg. 50% of the maximum value is recorded for use in the evaluation of proprioceptive strength sense. Then, isometric quadriceps femoris contraction is requested until the calculated proprioceptive force sense pressure value is reached. They are told to stay in this position for 5 seconds and then relax. Afterwards, individuals were asked to say when they thought they had reached this value without looking at the device screen. When the patients say "ok", the value on the screen is saved. The difference between this value and the calculated proprioceptive force sense value is recorded in mmHg. Measurements are repeated 3 times and the average is considered as the test result.

Lower Extremity Length Measurement: It is performed in order to compare the changes in the bone structure with the other side. Measurements are made with an inelastic tape measure. The patients to be measured are placed in the supine position. The distance between the trochanter major and the medial malleolus will be used for lower extremity length measurement. Measurements will be recorded in centimeters.

Lower Extremity Joint Range of Motion: One of the methods used to evaluate the joint range of motion in the clinic is the measurement made with the help of a goniometer.

WOMAC (Western Ontario-Macmaster Osteoarthritis Score): It is used to evaluate the functional status of patients with coxarthrosis and gonarthrosis. The validity and reliability of the test was done by Tuzun et al. It evaluates disability due to osteoarthritis. It consists of 3 parts: pain, stiffness and loss of physical function.

10 Meter Walking Test: It is a test used to evaluate walking speed. The first 3 and the last 3 meters of the created 16-meter track are not included in the time calculation. Time starts when the patient's first foot crosses the starting line, and ends when the second foot crosses the finish line. Three repetitions are performed and the average is taken. Evaluation will be performed by allowing adequate rest intervals between repetitions.

Tibiofemoral angle: It is calculated by AP X-ray taken while the patient is in the standing position. It is found by the angle between the anatomical axis of the femur and the anatomical axis of the tibia. Its normal value is between 2.20 and 7.40. This angle is affected by all angle-related values of the lower extremity. It is highly correlated with functional capacity. An angle above the normal value indicates valgus, and a decrease below the normal value indicates varus deformity in the lower extremity.

Knee medial compartment distance: The minimum width remaining medially between the tibia and the femur will be recorded in millimeters. The minimum joint space width will be measured as the distance between the bones in the medial tibiofemoral region. The minimum distance is between the distal femur and the proximal tibia. The point where the convex line of the medial condyle of the femur is lowest is marked. From this point, the place where the perpendicular drawn on the ground intersects with the tibial plateau is marked. The medial compartment distance of the knee is calculated by recording the distance in millimeters between these two marked points. The decrease in the distance can be interpreted as an increase in the varus deformity of the knee.

KOOS (Knee Injury and Osteoarthritis Outcome Score): It is used to evaluate the symptoms and functional status of knee OA. It consists of 5 subgroups. These are pain, activities of daily living, functional status in sports and leisure activities, knee-related quality of life. It consists of 42 questions in total. Each subscale is scored between 0 and 100 points.

SF-36: It is a scale used to evaluate quality of life. Turkish validity and reliability studies were conducted. The scale consists of 36 questions. It is divided into its own subheadings and used to measure the functional status of the person. It consists of eight parts. These sections are: social competence, cognitive health status, physical competence, pain, emotional strength, energy, general health perception, and physical strength. These parameters have different ratings. The scale is scored between 0 and 100 points in total. An increase in the score is interpreted as an improvement in health status.

Berg Balance Scale: It is used to evaluate both static and dynamic balance. It is a scale with Turkish validity and reliability. It consists of 14 items used in ADLs with increasing difficulty levels. The scoring of each item is between 0 and 4. The lowest score is 0 points and the highest 56 points. A score of 45 and above indicates good balance.

Tampa Kinesiophobia Scale (TKS) is a 17-item scale developed to measure fear of movement/re-injury. The scale includes the parameters of injury/re-injury and fear-avoidance in work-related activities. Turkish adaptation study Tunca Yılmaz Ö. carried out by et al. 4-point Likert scoring on the scale (1 = I strongly disagree, 4 = Totally I agree) is used. After reversing items 4, 8, 12 and 16, a total score is calculated. The person gets a total score between 17-68.

USG: Pennation angle calculation and muscle thickness measurement will be performed at the 4 heads of the Quadriceps Femoris muscle (vastus medialis, lateralis, intermedius and rectus femoris) before and after the treatment. These measurements will be evaluated from the middle of the thigh (between the trochanter major of the femur and the midpoint of the lateral condyle of the femur) while the patient is lying in the supine position. Muscle thickness will be measured as the distance between the superficial and deep aponeuroses by applying the vertical and maximum pressure of the USG probe.

Baseline Digital Inclinometer: It is used to evaluate joint position sense and range of motion in the clinic. It is a calibrated device with a margin of error of 1 degree. Position sense measurement knee extension For the right and left extremities, it will be done in the eyes open and eyes closed positions. The reposition angle method will be used in the measurement of joint position sense. According to this method; The patient's extremity is taken to the position where it should be taken by the physiotherapist. In this position, the patient is asked to remember this position by waiting for 5 seconds. In this position, the patient is asked to remember this position by waiting for 5 seconds. The patient is then asked to return the extremity to that position. In the measurement of knee extension, the inclinometer is fixed on the tibia while the patient sits on the side of the bed with their knees flexed at 90 degrees. From the position of the patient; 30 degrees and 60 degrees knee extension is requested. 3 repetitions are taken and the average is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 40-65,
* Those diagnosed with medial compartment knee OA, grade 2-3 according to the Kellgren-Lawrence classification,
* Patients who can stand on one leg for at least 30 seconds

Exclusion Criteria:

* Presence of neurological problems,
* Operation in the lower extremities or spinal column,
* Severe vision, speech, hearing problems,
* Inability to walk independently,
* Having a BMI of more than 35,
* Receiving physical therapy and rehabilitation due to gonarthrosis in the last year.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Muscle Architectural Evaluation with USG | 2 months
  Before and after the treatment, pennation angle calculation and muscle thickness measurement will be made at the 4 heads of the Quadriceps Femoris muscle (vastus medialis, lateralis, intermedius and rectus femoris). These measurements will be evaluated from the middle of the thigh (between the trochanter major of the femur and the midpoint of the lateral condyle of the femur) while the patient is lying in the supine position. Muscle thickness will be measured as the distance between the superficial and deep aponeuroses by applying the vertical and maximum pressure of the USG probe. Pennation angle measurement will be determined by placing the USG probe longitudinally from the middle of the thigh and measuring the angles where the muscle fascicles attach to the deep aponeurosis.
Knee medial compartment distance | 2 months
  The minimum width remaining medially between the tibia and the femur will be recorded in millimeters. The minimum joint space width will be measured as the distance between the bones in the medial tibiofemoral region. The minimum distance is between the distal femur and the proximal tibia. The point where the convex line of the medial condyle of the femur is lowest is marked. From this point, the place where the perpendicular drawn on the ground intersects with the tibial plateau is marked. The medial compartment distance of the knee is calculated by recording the distance in millimeters between these two marked points. The decrease in the distance can be interpreted as an increase in the varus deformity of the knee.
Tibiofemoral angle measurement | 2 months
  It is calculated by AP X-ray taken while the patient is in the standing position. It is found by the angle between the anatomical axis of the femur and the anatomical axis of the tibia. Its normal value is between 2.2 and 7.4. This angle is affected by all angle-related values of the lower extremity. Therefore, it is highly correlated with functional capacity. An angle above the normal value indicates valgus, and a decrease below the normal value indicates varus deformity in the lower extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih ERBAHÇECİ, Study Director — Hacettepe University; Eren ARABACI, Study Director — Amasya University
Locations (1):
- Amasya Healthy Life Center, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If deemed necessary, sharing will be made in case of need. Personal information will not be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 01.06.2023-01.16.2024
Access Criteria: Must be one of the researchers of this study

REFERENCES:
- [Background] Barrios JA, Higginson JS, Royer TD, Davis IS. Static and dynamic correlates of the knee adduction moment in healthy knees ranging from normal to varus-aligned. Clin Biomech (Bristol). 2009 Dec;24(10):850-4. doi: 10.1016/j.clinbiomech.2009.07.016. Epub 2009 Aug 22. PMID 19703728
- [Background] Lawrence RC, Helmick CG, Arnett FC, Deyo RA, Felson DT, Giannini EH, Heyse SP, Hirsch R, Hochberg MC, Hunder GG, Liang MH, Pillemer SR, Steen VD, Wolfe F. Estimates of the prevalence of arthritis and selected musculoskeletal disorders in the United States. Arthritis Rheum. 1998 May;41(5):778-99. doi: 10.1002/1529-0131(199805)41:53.0.CO;2-V. PMID 9588729
- [Background] Hunt MA, Birmingham TB, Bryant D, Jones I, Giffin JR, Jenkyn TR, Vandervoort AA. Lateral trunk lean explains variation in dynamic knee joint load in patients with medial compartment knee osteoarthritis. Osteoarthritis Cartilage. 2008 May;16(5):591-9. doi: 10.1016/j.joca.2007.10.017. Epub 2008 Feb 21. PMID 18206395
- [Background] Lephart SM, Pincivero DM, Rozzi SL. Proprioception of the ankle and knee. Sports Med. 1998 Mar;25(3):149-55. doi: 10.2165/00007256-199825030-00002. PMID 9554026
- [Background] Gellhorn AC, Stumph JM, Zikry HE, Creelman CA, Welbel R. Ultrasound measures of muscle thickness may be superior to strength testing in adults with knee osteoarthritis: a cross-sectional study. BMC Musculoskelet Disord. 2018 Sep 27;19(1):350. doi: 10.1186/s12891-018-2267-4. PMID 30261863